CLINICAL TRIAL: NCT04587544
Title: Effect of a Cold Water Immersion (CWI) on Pain in People With Gouty Arthritis: A Community Based Randomized Controlled Trial
Brief Title: The Relationship Between Cold Water Immersion and the Progression in Gout Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Maria Dyah Kurniasari, College of Nursing, Taipei Medical University, Taipei, Taiwan, R.O.C., Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N201912052
Record Dates: First submitted 2020-09-24; First posted 2020-10-14 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Gout Arthritis
Keywords: Gout Arthritis; Cold Water Immersion; Pain
MeSH Terms: conditions — Arthritis, Gouty; Pain

STUDY DESIGN:
Intervention Model Description: The randomized control trial study with two parallel-intervention-groups was employed to examine the effect of CWI (20-30C) therapy. All participants were randomly assigned to either CWI (20-30C) therapy intervention group or the control group. Block random sampling was then employed to generate the intervention and control group sequence. All participants were assessed on their pain as the primary outcome, joint mobility, stress, anxiety, depression, QOL (included PCS and MCS), physical activity (MET-h/week) at three times points: before the intervention, 2nd and 4th-week of the intervention.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, it is only possible to blind the evaluator of the study. The evaluator is blinded the group division either treatment or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold Water Immersion (Experimental): The participants maintained their daily activities during the intervention. When daily activity ended, the intervention was begun. CWI therapy by immersed the whole part of inflamed target joints in the water at 20-30C for 20 minutes/day. The intervention was continued for four weeks. The researchers work together with the nurses of community health services to give the intervention.
  Interventions: Behavioral: Cold Water Immersion
- No Intervention (No Intervention): The participants would not receive Cold Water Intervention. However, they are allowed to received the usual care

INTERVENTIONS:
Behavioral: Cold Water Immersion — The participants maintained their daily activities during the intervention. When daily activity ended, the intervention was begun. CWI therapy by immersed the whole part of inflamed target joints in the water at 20-30C for 20 minutes/day. The intervention was continued for four weeks. The researchers work together with the nurses of community health services to give the intervention.
  Arms: Cold Water Immersion

SUMMARY:
Gouty arthritis is a type of autoinflammatory arthritis that generates higher levels of pain with only minimum movement in the joint. The pain is shown to have a negative correlation with the physical function, reduced peak ankle joint angular, mobility velocity , and physical function. As such, the investigator can conclude that gout arthritis led to raises intolerance foot pain, physical inactivity, and joint mobility reduction. Currently, intermittent drugs use for pain relief is suggested to contribute to the renal impairment side effect. However, the investigator found that there is a limited study that investigated non-pharmacological intervention among people with gouty arthritis. The pain among people with gouty arthritis has also been shown to increase the degree of depression, anxiety, and depression. Also, the high levels of pain, psychological distress, anxiety, and depression were found as the risk factor of poor Quality of Life (QOL). Cold therapy (cryotherapy) application has been proven as useful adjuvant therapy on pain among people with gouty arthritis. CWI therapy has twofold reduced the inflammation. Firstly, it attenuates metabolic processes in stressed tissues and slowing cytokine and myokine up-regulation that mediates inflammation. Second, CWI induces microvasculature vasoconstriction by perfusing stressed tissue and reducing the circulatory of tissue access to inflammatory cells. Meanwhile, the high prevalence of gouty arthritis has been presented in North Celebes, Indonesia. Moreover, more than 50% of patients are too late for effective therapy and they had observed tophi for 7 to 9 years before presenting for treatment. These empirical issues indicate that it is vital to investigate gouty arthritis-related risk factors to protect Indonesians from this disease. The investigator aims to investigate a unique analysis of the CWI (20-30C) therapy effect on pain, joint mobility, stress, anxiety, depression, QOL (encompasses PCS and MCS), physical activity (MET-h/week) in the multicenter-community setting with a longitudinal study design.

DETAILED DESCRIPTION:
This research was conducted at North Celebes, Indonesia. Participants were recruited using the multi-stage sampling method, which began in July 2019. North Celebes Province was conveniently selected in the first stage sampling, which had the highest prevalence of gouty arthritis. North Celebes province is stratified it into 15 regions. In the second stage, two regions of fifteen regions were randomly selected, including urban and rural areas. Tomohon City is the one urban area that has been able to engage in this partnership. Seven Community Health Service (CHS) centers in Tomohon City have been randomly chosen in the final level. Four qualified professional nurses collected all the data. The data source of diagnoses was their medical records in the Public Community Health Services (CHS) of Tomohon City. The sample calculation utilized G-Power 3.1 software with the alpha level (α) of 0.01, power (1-ß) of 0.80, and the effect size is 0.9, the total estimated sample size required 31 in each group. An estimated 20% dropout rate increases; the sample size is 36 for each group.

Variable description 1.1.1. Participants Characteristic Blood pressure and BMI were examined in a standardized medical examination. Demographic data were collected by using a self-designed questionnaire. The questionnaire included the demographic characteristics of the participant, including age, gender, marital status, educational level, income, occupation, family gout history, gouty arthritis drug consumption, alcohol consumption, and smoking status. The translated food frequency questionnaire was employed with Cronbach's alpha as 0.95.

1.1.2. Pain The Visual Analog Scale (VAS) instrument has 10 centimeters length. The standard scale anchored by "no pain" marked as a score of 0 and the "worst imaginable pain" marked as a score of 10 cm. The higher score identifies greater pain intensity. The reliability test showed that VAS was good (r = 0.94, p = 0.001). The reliability test of the VAS instrument has been done in Indonesia with the Cronbach's alpha as 0.89.

1.1.3. Joint mobility The range of knee joint motion was calculated using an International Standard Orthopedic Measurement (ISOM) goniometric. Its method using the Sagittal Frontal Transverse Rotation (SFTR) system to an accuracy of 10. Goniometry provides an objective assessment tool to measure the range of motion. The validity and reliability of Goniometry are 0.98 and 0.97, respectively. The validity score of the Indonesian version is 0.97, and the Cronbach alpha as 0.51.

1.1.4. Stress, anxiety, depression The Depression Anxiety Stress Scale (DASS-21) questionnaire is used to measure the negative states of three mental health conditions: depression, anxiety, and stress using a self-report 4-point Likert scale. Data was collected by reflects the thoughts, feelings, and behavior. The result will be defined by the total scores of responses from the 7-item subscale of this questionnaire. The Cronbach's alphas of Indonesian translated is 0.72 to 0.87.

1.1.5. Quality of Life (QOL) 36 Health Survey (SF-36) questionnaire was employed to estimate QOL. It included Physical Component Summary (PCS), Mental Component Summary (MCS). Total QOL range from 0 to 100. The Indonesia version of the SF-36 questionnaire has tested the reliability with the Cronbach's alphas 0.7.

1.1.6. Physical activity (MET-h/week) The physical activity level was investigated as metabolic equivalent of task (MET)-hr/week by using three questions based on the modified Physical Activity Guideline from the Advisory Committee for Americans and the Godin Leisure-Time Exercise Questionnaire. The investigator then categorized participants based on the exercise type (that is divided into the following categories: mild (e.g., yoga, bowling, or floor-sweeping), moderate (e.g., gym, baseball, or badminton), and strenuous exercise (e.g., hiking, soccer, or running)), duration in minutes and exercise intensity they presented during a typical week. The investigator multiplied the amount of mild, moderate, and strenuous exercise hours and duration by 3, 5, and 9, respectively. By summing the exercise pattern of the separate things, the investigator measured total weekly PA in arbitrary units.

The per-protocol method was employed to deal with the missing data. Each participant is allowed to immediately report the adverse event during the intervention.

The Chi-square and t-test were employed to analyze the homogeneity of subject characteristics between the experimental and control group. The Generalized Estimating Equation (GEE) model was applied to compare the differences pain, joint mobility, stress, anxiety, depression, QOL (included PCS and MCS), physical activity (MET-h/week) within one-month intervention between the intervention and control group. The interaction between group and time was also further analyzed to determine if the mean differences in their pain, joint mobility, stress anxiety, and depression, QOL, and physical activity between groups differed significantly over time. p<0.05 was applied as statistically significant. All statistical analyses were performed using the Statistical Package for the Social Sciences (SPSS) vers. 25.0 (Chicago, IL, USA). Besides, Structural Equation Modeling (SEM) was also employed to analyze the mediating effect between variables through the Analysis of Moment Structures (AMOS) vers. 24. Then the investigator evaluate the measurement and structural models by utilizing the goodness fit index.

ELIGIBILITY:
Inclusion Criteria:

* People with gouty arthritis in the knee or ankle or metatarsophalangeal or metacarpophalangeal or olecranon bursa or wrist
* Participants were Indonesian nationals aged ≥18 years
* They had visited a clinic of the Public CHS of Tomohon City
* They had agreed to participate in the study.

Exclusion Criteria:

* Participants who self-reported the presence of other types of inflammatory arthritis, including RA or spondyloarthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Pain Level assessed by The Visual Analog Scale (VAS) at the baseline | Baseline/ pre-intervention
  Pain Level assessed by the Visual Analog Scale (VAS) instrument that has 10 centimeters length. The standard scale anchored by "no pain" marked as a score of 0 and the "worst imaginable pain" marked as a score of 10 cm (Huskisson et al., 1974; Scott & Huskisson, 1976). The higher score identifies greater pain intensity. The reliability test showed that VAS was good (r = 0.94, p = 0.001) (Ferraz et al., 1990). The reliability test of the VAS instrument has been done in Indonesia with the Cronbach's alpha as 0.89 (Suwendar et al., 2017)
Pain Level assessed by The Visual Analog Scale (VAS) at the 2nd week/during the intervention | 2nd week/during the intervention
  Pain Level assessed by The Visual Analog Scale (VAS) instrument that has 10 centimeters length. The standard scale anchored by "no pain" marked as a score of 0 and the "worst imaginable pain" marked as a score of 10 cm (Huskisson et al., 1974; Scott & Huskisson, 1976). The higher score identifies greater pain intensity. The reliability test showed that VAS was good (r = 0.94, p = 0.001) (Ferraz et al., 1990). The reliability test of the VAS instrument has been done in Indonesia with the Cronbach's alpha as 0.89 (Suwendar et al., 2017)
Pain Level assessed by the Visual Analog Scale (VAS) at 4th week/immediately after intervention | 4th week/immediately after intervention
  Pain Level assessed by the Visual Analog Scale (VAS) instrument has 10 centimeters length. The standard scale anchored by "no pain" marked as a score of 0 and the "worst imaginable pain" marked as a score of 10 cm (Huskisson et al., 1974; Scott & Huskisson, 1976). The higher score identifies greater pain intensity. The reliability test showed that VAS was good (r = 0.94, p = 0.001) (Ferraz et al., 1990). The reliability test of the VAS instrument has been done in Indonesia with the Cronbach's alpha as 0.89 (Suwendar et al., 2017)

SECONDARY OUTCOMES:
Joint mobility assessed by Goniometry at the baseline | Baseline/ pre-intervention
  Joint mobility assessed by Goniometry. The range of knee joint motion was calculated using an International Standard Orthopedic Measurement (ISOM) goniometric. Its method using the Sagittal Frontal Transverse Rotation (SFTR) system to an accuracy of 10 (Dorwart, Hansell, & Schumacher, 1974). Goniometry provides an objective assessment tool to measure the range of motion (Rose & Norton, 1987). The validity and reliability of Goniometry are 0.98 and 0.97, respectively (Rose & Norton, 1987). The validity score of the Indonesian version is 0.97, and the Cronbach alpha as 0.51 (Hafiyah, 2013).
Joint mobility assessed by Goniometry at the 2nd week/during the intervention | 2nd week/during the intervention
  Joint mobility assessed by Goniometry. The range of knee joint motion was calculated using an International Standard Orthopedic Measurement (ISOM) goniometric. Its method using the Sagittal Frontal Transverse Rotation (SFTR) system to an accuracy of 10 (Dorwart, Hansell, & Schumacher, 1974). Goniometry provides an objective assessment tool to measure the range of motion (Rose & Norton, 1987). The validity and reliability of Goniometry are 0.98 and 0.97, respectively (Rose & Norton, 1987). The validity score of the Indonesian version is 0.97, and the Cronbach alpha as 0.51 (Hafiyah, 2013).
Joint mobility assessed by Goniometry at the 4th week/immediately after intervention | 4th week/immediately after intervention
  Joint mobility assessed by Goniometry. The range of knee joint motion was calculated using an International Standard Orthopedic Measurement (ISOM) goniometric. Its method using the Sagittal Frontal Transverse Rotation (SFTR) system to an accuracy of 10 (Dorwart, Hansell, & Schumacher, 1974). Goniometry provides an objective assessment tool to measure the range of motion (Rose & Norton, 1987). The validity and reliability of Goniometry are 0.98 and 0.97, respectively (Rose & Norton, 1987). The validity score of the Indonesian version is 0.97, and the Cronbach alpha as 0.51 (Hafiyah, 2013).
Stress, anxiety, depression assessed by The Depression Anxiety Stress Scale questionnaire at the baseline | Baseline/ pre-intervention
  The Depression Anxiety Stress Scale questionnaire is used to measure the negative states of three mental health conditions: depression, anxiety, and stress using a self-report 4-point Likert scale. Data was collected by reflects the thoughts, feelings, and behavior (Oei, Sawang, Goh, & Mukhtar, 2013). The result will be defined by the total scores of responses from the 7-item subscale of this questionnaire. The lower score shows a better result. If the total number of depressions is 9 or below and the extremely severe is 34 or over. The Cronbach's alphas of Indonesian translated is 0.72 to 0.87 (Susilowati, Isahak, & Harncharoen, 2016).
Stress, anxiety, depression assessed by The Depression Anxiety Stress Scale questionnaire at the 2nd week/during the intervention | 2nd week/during the intervention
  The Depression Anxiety Stress Scale questionnaire is used to measure the negative states of three mental health conditions: depression, anxiety, and stress using a self-report 4-point Likert scale. Data was collected by reflects the thoughts, feelings, and behavior (Oei, Sawang, Goh, & Mukhtar, 2013). The result will be defined by the total scores of responses from the 7-item subscale of this questionnaire. The lower score shows a better result. If the total number of depressions is 9 or below and the extremely severe is 34 or over. The Cronbach's alphas of Indonesian translated is 0.72 to 0.87 (Susilowati, Isahak, & Harncharoen, 2016).
Stress, anxiety, depression assessed by the Depression Anxiety Stress Scale at 4th week/immediately after intervention | 4th week/immediately after intervention
  The Depression Anxiety Stress Scale questionnaire is used to measure the negative states of three mental health conditions: depression, anxiety, and stress using a self-report 4-point Likert scale. Data was collected by reflects the thoughts, feelings, and behavior (Oei, Sawang, Goh, & Mukhtar, 2013). The result will be defined by the total scores of responses from the 7-item subscale of this questionnaire. The lower score shows a better result. If the total number of depressions is 9 or below and the extremely severe is 34 or over. The Cronbach's alphas of Indonesian translated is 0.72 to 0.87 (Susilowati, Isahak, & Harncharoen, 2016).
Quality of Life (QOL) level assessed by 36 Health Survey (SF-36) questionnaire at Baseline | Baseline, pre-intervention
  Quality of Life (QOL) level assessed by 36 Health Survey (SF-36) questionnaire that was employed to estimate QOL. It included Physical Component Summary (PCS), Mental Component Summary (MCS). Total QOL range from 0 to 100 (Rias et al., 2020). The Indonesia version of the SF-36 questionnaire has tested the reliability with the Cronbach's alphas 0.7 (Salim, Yamin, Alwi, & Setiati, 2015)
Quality of Life (QOL) level assessed by 36 Health Survey (SF-36) questionnaire 2nd week/during the intervention | 2nd week/during the intervention
  Quality of Life (QOL) level assessed by 36 Health Survey (SF-36) questionnaire that was employed to estimate QOL. It included Physical Component Summary (PCS), Mental Component Summary (MCS). Total QOL range from 0 to 100 (Rias et al., 2020). The Indonesia version of the SF-36 questionnaire has tested the reliability with the Cronbach's alphas 0.7 (Salim, Yamin, Alwi, & Setiati, 2015)
Quality of Life (QOL) level assessed by36 Health Survey (SF-36) questionnaire 4th week/immediately after intervention | 4th week/immediately after intervention
  Quality of Life (QOL) level assessed by 36 Health Survey (SF-36) questionnaire that was employed to estimate QOL. It included Physical Component Summary (PCS), Mental Component Summary (MCS). Total QOL range from 0 to 100 (Rias et al., 2020). The Indonesia version of the SF-36 questionnaire has tested the reliability with the Cronbach's alphas 0.7 (Salim, Yamin, Alwi, & Setiati, 2015)
Physical activity (MET-h/week) level assessed by questions based on the modified Physical Activity Guideline at the baseline | Baseline, pre-intervention
  The physical activity level was investigated as metabolic equivalent of task (MET)-hr/week by using three questions based on the modified Physical Activity Guideline from the Advisory Committee for Americans (Shiroma, Sesso, Moorthy, Buring, & Lee, 2015) and the Godin Leisure-Time Exercise Questionnaire (Godin & Shephard, 1997). We then categorized participants based on the exercise type (that is divided into the following categories: mild (e.g., yoga, bowling, or floor-sweeping), moderate (e.g., gym, baseball, or badminton), and strenuous exercise (e.g., hiking, soccer, or running)), duration in minutes and exercise intensity they presented during a typical week. We multiplied the amount of mild, moderate, and strenuous exercise hours and duration by 3, 5, and 9, respectively. By summing the exercise pattern of the separate things, we measured total weekly PA in arbitrary units (Rias et al., 2020).
Physical activity (MET-h/week) level assessed by questions based on the modified Physical Activity Guideline at 2nd week/during the intervention | 2nd week/during the intervention
  The physical activity level was investigated as metabolic equivalent of task (MET)-hr/week by using three questions based on the modified Physical Activity Guideline from the Advisory Committee for Americans (Shiroma, Sesso, Moorthy, Buring, & Lee, 2015) and the Godin Leisure-Time Exercise Questionnaire (Godin & Shephard, 1997). We then categorized participants based on the exercise type (that is divided into the following categories: mild (e.g., yoga, bowling, or floor-sweeping), moderate (e.g., gym, baseball, or badminton), and strenuous exercise (e.g., hiking, soccer, or running)), duration in minutes and exercise intensity they presented during a typical week. We multiplied the amount of mild, moderate, and strenuous exercise hours and duration by 3, 5, and 9, respectively. By summing the exercise pattern of the separate things, we measured total weekly PA in arbitrary units (Rias et al., 2020).
Physical activity (MET-h/week) level: Change from Baseline and 2nd week time point | 4th week/immediately after intervention
  The physical activity level was investigated as metabolic equivalent of task (MET)-hr/week by using three questions based on the modified Physical Activity Guideline from the Advisory Committee for Americans (Shiroma, Sesso, Moorthy, Buring, & Lee, 2015) and the Godin Leisure-Time Exercise Questionnaire (Godin & Shephard, 1997). We then categorized participants based on the exercise type (that is divided into the following categories: mild (e.g., yoga, bowling, or floor-sweeping), moderate (e.g., gym, baseball, or badminton), and strenuous exercise (e.g., hiking, soccer, or running)), duration in minutes and exercise intensity they presented during a typical week. We multiplied the amount of mild, moderate, and strenuous exercise hours and duration by 3, 5, and 9, respectively. By summing the exercise pattern of the separate things, we measured total weekly PA in arbitrary units (Rias et al., 2020).

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu Ting Tsai, PhD, Study Director — Taipei Medical University
Locations (1):
- Rendra, Tomohon, North Celebes, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abhishek A, Doherty M. Education and non-pharmacological approaches for gout. Rheumatology (Oxford). 2018 Jan 1;57(suppl_1):i51-i58. doi: 10.1093/rheumatology/kex421. PMID 29272507
- [Background] Bleakley C, McDonough S, Gardner E, Baxter GD, Hopkins JT, Davison GW. Cold-water immersion (cryotherapy) for preventing and treating muscle soreness after exercise. Cochrane Database Syst Rev. 2012 Feb 15;2012(2):CD008262. doi: 10.1002/14651858.CD008262.pub2. PMID 22336838
- [Background] Burke BT, Kottgen A, Law A, Windham BG, Segev D, Baer AN, Coresh J, McAdams-DeMarco MA. Physical Function, Hyperuricemia, and Gout in Older Adults. Arthritis Care Res (Hoboken). 2015 Dec;67(12):1730-8. doi: 10.1002/acr.22648. PMID 26138016
- [Background] Albar, Z. (2007). Gout: Diagnosis and management. Medical Journal of Indonesia, 16(1), 47-54. https://doi.org/10.13181/mji.v16i1.256
- [Background] Amanah, A., Komala, I., Kurniasari, M. D., Dharmana, E., & Gasem, M. H. (2018). Effect of Mangosteen ( Garcinia mangostana ) PEEL Extract towards CD4 + , CD8 + T LYMPHOCYTES , CD38 Expression , NK Cells , IL-2 and IFN γ in Hiv Patients with Antiretroviral Therapy. Hiroshima Journal of Medical Sciences, 67(24), 56-62.
- [Background] Carroll M, Boocock M, Dalbeth N, Stewart S, Frampton C, Rome K. Ankle joint function during walking in tophaceous gout: A biomechanical gait analysis study. Gait Posture. 2018 Jun;63:150-153. doi: 10.1016/j.gaitpost.2018.04.020. Epub 2018 Apr 17. PMID 29734124
- [Background] Chandratre P, Mallen CD, Roddy E, Liddle J, Richardson J. "You want to get on with the rest of your life": a qualitative study of health-related quality of life in gout. Clin Rheumatol. 2016 May;35(5):1197-205. doi: 10.1007/s10067-015-3039-2. Epub 2015 Aug 6. PMID 26245722
- [Background] Chandratre P, Mallen C, Richardson J, Muller S, Hider S, Rome K, Blagojevic-Bucknall M, Roddy E. Health-related quality of life in gout in primary care: Baseline findings from a cohort study. Semin Arthritis Rheum. 2018 Aug;48(1):61-69. doi: 10.1016/j.semarthrit.2017.12.005. Epub 2018 Jan 5. PMID 29398125
- [Background] DiBonaventura Md, Andrews LM, Yadao AM, Kahler KH. The effect of gout on health-related quality of life, work productivity, resource use and clinical outcomes among patients with hypertension. Expert Rev Pharmacoecon Outcomes Res. 2012 Dec;12(6):821-9. doi: 10.1586/erp.12.60. PMID 23252362
- [Background] Dorwart BB, Hansell JR, Schumacher HR Jr. Effects of cold and heat on urate crystal-induced synovitis in the dog. Arthritis Rheum. 1974 Sep-Oct;17(5):563-71. doi: 10.1002/art.1780170510. No abstract available. PMID 4413123
- [Background] Ferraz MB, Quaresma MR, Aquino LR, Atra E, Tugwell P, Goldsmith CH. Reliability of pain scales in the assessment of literate and illiterate patients with rheumatoid arthritis. J Rheumatol. 1990 Aug;17(8):1022-4. PMID 2213777
- [Background] Fields TR. The Challenges of Approaching and Managing Gout. Rheum Dis Clin North Am. 2019 Feb;45(1):145-157. doi: 10.1016/j.rdc.2018.09.009. PMID 30447743
- [Background] Fu T, Cao H, Yin R, Zhang L, Zhang Q, Li L, Gu Z. Associated factors with functional disability and health-related quality of life in Chinese patients with gout: a case-control study. BMC Musculoskelet Disord. 2017 Nov 3;18(1):429. doi: 10.1186/s12891-017-1787-7. PMID 29100504
- [Background] Godin, G., & Shephard, R. J. . (1997). Godin leisure-time exercise questionnaire. Medicine and Science in Sports and Exercise, 29(6), 36-38.
- [Background] Hafiyah, F. (2013). Kontribusi Fleksibilitas Pergelangan Tangan dan Fleksibilitas Pinggang Terhadap Hasil Standing Shoot Dalam Perainan Bola Tangan Jurnal. Bandung.
- [Background] Hair, J. F., Ringle, C. M., Sarstedt, M., Hair, J. F., Ringle, C. M., & Sarstedt, M. (2014). PLS-SEM : Indeed a Silver Bullet. Journal of Marketing Theory and Practice, 19(2), 37-41. https://doi.org/10.2753/MTP1069-6679190202
- [Background] Harth M, Nielson WR. Pain and affective distress in arthritis: relationship to immunity and inflammation. Expert Rev Clin Immunol. 2019 May;15(5):541-552. doi: 10.1080/1744666X.2019.1573675. Epub 2019 Feb 11. PMID 30669892
- [Background] Health Research and Development Agency. (2013). Riset Kesehatan Dasar (RISKESDAS) 2013. Laporan Nasional 2013, 1-384. https://doi.org/1 Desember 2013
- [Background] Hilderink PH, Burger H, Deeg DJ, Beekman AT, Oude Voshaar RC. The temporal relation between pain and depression: results from the longitudinal aging study Amsterdam. Psychosom Med. 2012 Nov-Dec;74(9):945-51. doi: 10.1097/PSY.0b013e3182733fdd. Epub 2012 Oct 31. PMID 23115345
- [Background] Hirsch JD, Terkeltaub R, Khanna D, Singh J, Sarkin A, Shieh M, Kavanaugh A, Lee SJ. Gout disease-specific quality of life and the association with gout characteristics. Patient Relat Outcome Meas. 2010 Mar 1;2010:1-8. doi: 10.2147/PROM.S8310. PMID 21686040
- [Background] Huskisson EC, Wojtulewski JA, Berry H, Scott J, Hart FD, Balme HW. Treatment of rheumatoid arthritis with fenoprofen: comparison with aspirin. Br Med J. 1974 Feb 2;1(5900):176-80. doi: 10.1136/bmj.1.5900.176. PMID 4590669
- [Background] Jaliana, Suhadi, La Ode, M., & Sety. (2018). The Related Factors With The Incidence of Uric Acid Among Patients Age 20-44 Years Old In Bahteramas General Hospital of Southest Sulawesi Province in 2017. Jurnal Ilmiah Mahasiswa Kesehatan Masyarakat, 3(2), 1-13.
- [Background] Jastrzabek R, Straburzynska-Lupa A, Rutkowski R, Romanowski W. Effects of different local cryotherapies on systemic levels of TNF-alpha, IL-6, and clinical parameters in active rheumatoid arthritis. Rheumatol Int. 2013 Aug;33(8):2053-60. doi: 10.1007/s00296-013-2692-5. Epub 2013 Feb 10. PMID 23397259
- [Background] Klich S, Krymski I, Michalik K, Kawczynski A. Effect of short-term cold-water immersion on muscle pain sensitivity in elite track cyclists. Phys Ther Sport. 2018 Jul;32:42-47. doi: 10.1016/j.ptsp.2018.04.022. Epub 2018 May 1. PMID 29738892
- [Background] Lin S, Zhang H, Ma A. Association of gout and depression: A systematic review and meta-analysis. Int J Geriatr Psychiatry. 2018 Mar;33(3):441-448. doi: 10.1002/gps.4789. Epub 2017 Sep 18. PMID 28921661
- [Background] Majumder, S. (2015). The village that just got its first fridge. BBC News, Calcutta. Retrieved from https://www.bbc.com/news/magazine-30925252
- [Background] Metzger D, Zwingmann C, Protz W, Jackel WH. [Whole-body cryotherapy in rehabilitation of patients with rheumatoid diseases--pilot study]. Rehabilitation (Stuttg). 2000 Apr;39(2):93-100. doi: 10.1055/s-2000-14442. German. PMID 10832164
- [Background] Nilawati, N. S., Nugraheni, S. A., & Frieda, N. (2005). Hubungan Konsumsi Ikan dengan Perkembangan Kognisi Anak Baduta (12 - 23 Bulan), Studi di Kecamatan Gandus Kota Palembang Tahun 2006. Jurnal Psikologi Universitas Gadjah Mada, 33(2), 1-6.
- [Background] Oei TP, Sawang S, Goh YW, Mukhtar F. Using the Depression Anxiety Stress Scale 21 (DASS-21) across cultures. Int J Psychol. 2013;48(6):1018-29. doi: 10.1080/00207594.2012.755535. Epub 2013 Feb 21. PMID 23425257
- [Background] Padang C, Muirden KD, Schumacher HR, Darmawan J, Nasution AR. Characteristics of chronic gout in Northern Sulawesi, Indonesia. J Rheumatol. 2006 Sep;33(9):1813-7. PMID 16960942
- [Background] Rhind SG, Castellani JW, Brenner IK, Shephard RJ, Zamecnik J, Montain SJ, Young AJ, Shek PN. Intracellular monocyte and serum cytokine expression is modulated by exhausting exercise and cold exposure. Am J Physiol Regul Integr Comp Physiol. 2001 Jul;281(1):R66-75. doi: 10.1152/ajpregu.2001.281.1.R66. PMID 11404280
- [Background] Rias YA, Kurniasari MD, Traynor V, Niu SF, Wiratama BS, Chang CW, Tsai HT. Synergistic Effect of Low Neutrophil-Lymphocyte Ratio With Physical Activity on Quality of Life in Type 2 Diabetes Mellitus: A Community-Based Study. Biol Res Nurs. 2020 Jul;22(3):378-387. doi: 10.1177/1099800420924126. Epub 2020 May 11. PMID 32390456
- [Background] Rock KL, Kataoka H, Lai JJ. Uric acid as a danger signal in gout and its comorbidities. Nat Rev Rheumatol. 2013 Jan;9(1):13-23. doi: 10.1038/nrrheum.2012.143. Epub 2012 Sep 4. PMID 22945591
- [Background] Gogia PP, Braatz JH, Rose SJ, Norton BJ. Reliability and validity of goniometric measurements at the knee. Phys Ther. 1987 Feb;67(2):192-5. doi: 10.1093/ptj/67.2.192. PMID 3809242
- [Background] Salim S, Yamin M, Alwi I, Setiati S. Validity and Reliability of the Indonesian Version of SF-36 Quality of Life Questionnaire on Patients with Permanent Pacemakers. Acta Med Indones. 2017 Jan;49(1):10-16. PMID 28450649
- [Background] Schlesinger N. Response to application of ice may help differentiate between gouty arthritis and other inflammatory arthritides. J Clin Rheumatol. 2006 Dec;12(6):275-6. doi: 10.1097/01.rhu.0000249864.95389.cf. PMID 17149056
- [Background] Schlesinger N, Detry MA, Holland BK, Baker DG, Beutler AM, Rull M, Hoffman BI, Schumacher HR Jr. Local ice therapy during bouts of acute gouty arthritis. J Rheumatol. 2002 Feb;29(2):331-4. PMID 11838852
- [Background] Scott J, Huskisson EC. Graphic representation of pain. Pain. 1976 Jun;2(2):175-84. No abstract available. PMID 1026900
- [Background] Shiroma EJ, Sesso HD, Moorthy MV, Buring JE, Lee IM. Do moderate-intensity and vigorous-intensity physical activities reduce mortality rates to the same extent? J Am Heart Assoc. 2014 Oct 17;3(5):e000802. doi: 10.1161/JAHA.114.000802. PMID 25326527
- [Background] Singh JA, Bharat A, Khanna D, Aquino-Beaton C, Persselin JE, Duffy E, Elashoff D, Khanna PP. Racial differences in health-related quality of life and functional ability in patients with gout. Rheumatology (Oxford). 2017 Jan;56(1):103-112. doi: 10.1093/rheumatology/kew356. Epub 2016 Oct 25. PMID 28028159
- [Background] Susilowati, I., Isahak, M., & Harncharoen, K. (2016). Depression, Anxiety and Stress among Small and Medium Enterprise Workers in Indonesia, Malaysia, Thailand, and Vietnam. International Journal Of Occupational Health and Public Health Nursing, 3(2), 13-29.
- [Background] Suwendar, S., Fudholi, A., Andayani, T. M., & Sastramihardja, H. S. (2017). Quality of Life Evaluation of Cervical Cancer Inpatients Before and After Chemotherapy by Using the EQ-5D Questionnaire. Indonesian Journal of Clinical Pharmacy, 6(1), 1-10. https://doi.org/10.15416/ijcp.2017.6.1.1
- [Background] Tsai HT, Tsai YM, Yang SF, Wu KY, Chuang HY, Wu TN, Ho CK, Lin CC, Kuo YS, Wu MT. Lifetime cigarette smoke and second-hand smoke and cervical intraepithelial neoplasm--a community-based case-control study. Gynecol Oncol. 2007 Apr;105(1):181-8. doi: 10.1016/j.ygyno.2006.11.012. Epub 2007 Jan 3. PMID 17204311
- [Background] Weinberger A, Fadilah R, Lev A, Pinkhas J. Intra-articular temperature measurements after superficial heating. Scand J Rehabil Med. 1989;21(1):55-7. PMID 2711138
- [Background] White G, Caterini JE. Cold water immersion mechanisms for recovery following exercise: cellular stress and inflammation require closer examination. J Physiol. 2017 Feb 1;595(3):631-632. doi: 10.1113/JP273659. No abstract available. PMID 28145015

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT04587544/Prot_SAP_ICF_000.pdf